CLINICAL TRIAL: NCT04642053
Title: A Randomized Control Trial of Motor-based Intervention for Childhood Apraxia of Speech
Brief Title: A Randomized Control Trial of Motor-based Intervention for CAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01DC018581-01 (NIH)
Record Dates: First submitted 2020-11-12; First posted 2020-11-24 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Childhood Apraxia of Speech
Keywords: Pediatric motor speech disorder; Speech motor control
MeSH Terms: conditions — Apraxias

STUDY DESIGN:
Intervention Model Description: This work will employ a delayed treatment control group design across multiple behaviors. Participants will be seen in two groups: an Immediate Treatment group and a Delayed Treatment group.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessors will be blind to treatment phase/session (i.e. Pre-Treatment, Treatment (including session #) and Maintenance), group (i.e. Immediate vs. Delayed) and word status (i.e. Treated vs. Untreated). They will performed blinded ratings of Word Accuracy and Speech Intelligibility, as well as blinded scoring of Duration and Variability.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Treatment (Experimental): Participants in the Immediate Treatment Group will receive DTTC Treatment four times per week (45-minute sessions each) for 8 weeks. Total duration will be 180 minutes/week over 32 sessions. Treatment will begin between 1-3 weeks following the diagnostic evaluation.
  Interventions: Behavioral: Dynamic Temporal and Tactile Cuing
- Delayed Treatment (Experimental): The Delayed Treatment Group serves as a control during the period in which participants are waiting to begin treatment. A delayed treatment onset is employed to control for maturation effects. Participants in the Delayed Treatment Group will receive DTTC Treatment four times per week (45-minute sessions each) for 8 weeks. Total duration will be 180 minutes/week over 32 sessions. Treatment will begin after an 8-week delay following the diagnostic evaluation.
  Interventions: Behavioral: Dynamic Temporal and Tactile Cuing

INTERVENTIONS:
Behavioral: Dynamic Temporal and Tactile Cuing — Dynamic Temporal and Tactile Cuing is based on principles of integral stimulation where the client watches, listens to and imitates the clinician (Strand, 2020). Treatment will begin by training the child to imitate and simultaneously produce syllables/words with the clinician. Sessions will focus on establishing accurate movement transitions in treated words. The child will be asked to imitate the clinician's production of the target. If the child's imitation is inaccurate, they will be instructed to simultaneously produce the target with the clinician. Simultaneous productions will continue to provide practice opportunity with maximal cuing. As the child gains greater accuracy, simultaneous productions will be faded and direct imitation will be attempted again. Over the course of treatment, the movement gesture will be shaped with the goal being accurate production with normal rate and naturalness.

SUMMARY:
Childhood apraxia of speech (CAS) is a complex, multivariate speech motor disorder characterized by difficulty planning and programming movements of the speech articulators (ASHA, 2007; Ayres, 1985; Campbell et al., 2007; Davis et al., 1998; Forrest, 2003; Shriberg et al., 1997). Despite the profound impact that CAS can have on a child's ability to communicate, little data are available to direct treatment in this challenging population. Historically, children with CAS have been treated with articulation and phonologically based approaches with limited effectiveness in improving speech, as shown by very slow treatment progress and poor generalization of skills to new contexts. With the emerging data regarding speech motor deficits in CAS, there is a critical need to test treatments that directly refine speech movements using methods that quantify speech motor control.

This research is a Randomized Control Trial designed to examine the outcomes of a non-traditional, motor-based approach, Dynamic Temporal and Tactile Cuing (DTTC), to improve speech production in children with CAS. The overall objectives of this research are (i) to test the efficacy of DTTC in young children with CAS (N=72) by examining the impact of DTTC on treated words, generalization to untreated words and post-treatment maintenance, and (ii) to examine how individual patterns of speech motor variability impact response to DTTC.

DETAILED DESCRIPTION:
Seventy-two children with CAS, between the ages of 2.5 and 7.11 years of age will be treated with DTTC. This work will employ a delayed treatment control group design across multiple behaviors. Participants will be seen in two groups: an Immediate Treatment group and a Delayed Treatment group. Probe data will be collected during the Pre-Treatment (5 data points), Treatment (12 data points) and Maintenance (minimum 5 data points) phases. The study duration is 28 weeks in total duration for all participants. The study will address the following specific aims:

Aim 1: Quantify the effects of DTTC on improved speech production (perceptual ratings) in treated words that are maintained post-treatment and generalized to untreated words in children with CAS. The working hypothesis is that DTTC will increase accuracy of treated words (primary outcome measure) and this effect will be maintained post-treatment and generalized to untreated words. We also predict that DTTC will increase speech intelligibility pre to post-treatment (secondary outcome measure).

Aim 2: Quantify the effects of DTTC on refined speech motor control (kinematic/acoustic measures) in treated words that are maintained post-treatment and generalized to untreated words in children with CAS. The working hypothesis is that DTTC will be associated with decreases in speech motor variability and duration of treated words (secondary outcome measures) that are maintained pre- to post-treatment and generalized to untreated words.

Aim 3: Characterize the effects of speech motor variability (within-subject) at baseline as a predictor of DTTC efficacy in children with CAS. The working hypothesis is that children with CAS who demonstrate higher levels of speech motor variability at baseline will display greater improvements in speech production accuracy following DTTC than children with lower levels of variability at baseline.

Treatment will be provided four times/week for 45-minute sessions. Principles of motor learning will be incorporated into sessions by controlling the type of practice (blocked vs. randomized), type of feedback (knowledge of results vs. knowledge of performance) and amount of feedback provided.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of childhood apraxia of speech (CAS). Diagnostic classification for CAS will be determined according to the presence of the three core features identified in the ASHA position statement on CAS: 1) inconsistent consonant and vowel errors over productions of repeated trials; 2) difficulties forming accurate movement between sounds and syllables; and 3) prosodic errors (ASHA, 2007). These three characteristics must be present in more than one speaking context (i.e. single words, connected speech, sequencing tasks). In addition to the three core features, children with CAS must demonstrate at least four of the following characteristics: vowel errors, timing errors, phoneme distortions, articulatory groping, impaired volitional oral movement, reduced phonetic inventory and poorer expressive than receptive language skills, which is consistent with the Strand 10-point checklist (Shriberg et al., 2012). We will identify the presence of these factors from the Dynamic Evaluation of Motor Speech Skills (DEMSS, Strand et al., 2013), Verbal Motor Production Assessment for Children (VMPAC, Hayden & Square, 1999), Goldman Fristoe Test of Articulation (GFTA-3, Goldman & Fristoe, 2016), and a connected speech sample. We have used these stringent criteria for diagnosing CAS in our past research (Please see the Diagnostic Framework and Criteria for CAS in Grigos and Case (2017)). The diagnosis will be made independently by two speech language pathologists (one being the PI) with expertise in assessing and treating children with CAS.
2. Age between 2.5 and 7.11 years of age.
3. Normal structure of the oral-peripheral mechanism.
4. Participants must pass a hearing screening conducted at 20 dB SPL at 500, 1000, 2000 and 4000 Hz.
5. No prior DTTC treatment.

Exclusion Criteria:

1. Positive history of neurological disorder (e.g. cerebral palsy), developmental disorder (e.g. autism spectrum disorder) or genetic disorder (e.g. Down syndrome).
2. Characteristics of dysarthria, even if the child meets criteria for CAS.
3. Fluency disorder, even if the child meets criteria for CAS.
4. Conductive or sensorineural hearing loss, even if the child meets criteria for CAS.
5. History of DTTC treatment.

Ages: 29 Months to 95 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Estimated)
Dates: Start 2021-09-14 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Changes in word accuracy | Through the treatment phase (32 treatment sessions over 8 weeks)
  Word accuracy will be quantified for treated and untreated words using a composite score that reflects accuracy of segmental and suprasegmental components of words.

SECONDARY OUTCOMES:
Changes in the percentage of words correctly identified by a listener | Pre to post-treatment (8-weeks from treatment onset)
  Standard procedures (Hustad et al., 2007; 2016) will be used to measure speech intelligibility by computing the percentage of intelligible words (treated and untreated). Five naïve adult listeners will orthographically transcribe randomized word productions from each child.
Changes in the speech motor variability of segments and words | Pre to post-treatment (8-weeks from treatment onset)
  Variability will be measured using acoustic and kinematic methods. Acoustic measures will include coefficient of variation of word and segment duration. Kinematic measures will include lip and jaw movement variability associated with whole word productions (i.e. spatiotemporal index (STI, Smith et al.1995) and coefficient of variation of single movements (i.e. movement from oral closing into oral opening; movement from oral opening into oral closing).
Changes in the duration of segments and words | Pre to post-treatment (8-weeks from treatment onset)
  Word and segment duration will be measured using acoustic and kinematic methods. Acoustic measures will include word and segment duration. Kinematic measures will include word and single movement duration (e.g. oral opening into vowel).

CONTACTS AND LOCATIONS:
Overall Officials: Maria I Grigos, PhD, Principal Investigator — New York University
Locations (1):
- New York University, Department of Communicative Sciences & Disordesr, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data tied to the primary and secondary outcome measures will be shared after deidentification.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 6 months following publication. No end date.
Access Criteria: Researchers and speech language pathologists who provide a methodologically sound proposal. Proposals should be directed to maria.grigos@nyu.edu. To gain access, data requestors will need to complete and sign a data sharing agreement.

REFERENCES:
- [Background] American Speech-Language-Hearing Association (2007). Childhood apraxia of speech: Technical Report. Available online: https://www.asha.org/policy/tr2007-00278/
- [Background] Ayres, A. J. (1985). Developmental dyspraxia and adult-onset apraxia: By A. Jean Ayres. Sensory integration international.
- [Background] Campbell TF, Dollaghan CA, Rockette HE, Paradise JL, Feldman HM, Shriberg LD, Sabo DL, Kurs-Lasky M. Risk factors for speech delay of unknown origin in 3-year-old children. Child Dev. 2003 Mar-Apr;74(2):346-57. doi: 10.1111/1467-8624.7402002. PMID 12705559
- [Background] Davis, B. L., Jakielski, K. J., & Marquardt, T. P. (1998). Developmental apraxia of speech: Determiners of differential diagnosis. Clinical Linguistics & Phonetics, 12(1), 25-45.
- [Background] Forrest K. Diagnostic criteria of developmental apraxia of speech used by clinical speech-language pathologists. Am J Speech Lang Pathol. 2003 Aug;12(3):376-80. doi: 10.1044/1058-0360(2003/083). PMID 12971826
- [Background] Goldman, R. & Fristoe, M. (2016). Goldman Fristoe Test of Articulation - 3. Circle Pines, MN: American Guidance Service
- [Background] Grigos MI, Case J. Changes in movement transitions across a practice period in childhood apraxia of speech. Clin Linguist Phon. 2018;32(7):661-687. doi: 10.1080/02699206.2017.1419378. Epub 2017 Dec 27. PMID 29281317
- [Background] Hayden, D. A., & Square, P. A. (1999). VMPAC: Verbal Motor Production Assessment for Children. San Antonio, TX: Psychological Association.
- [Background] Hustad KC, Allison KM, Sakash A, McFadd E, Broman AT, Rathouz PJ. Longitudinal development of communication in children with cerebral palsy between 24 and 53 months: Predicting speech outcomes. Dev Neurorehabil. 2017 Aug;20(6):323-330. doi: 10.1080/17518423.2016.1239135. Epub 2016 Oct 28. PMID 27792399
- [Background] Hustad, K. C. and Weismer,G. (2007). A continuum of interventions for individuals with dysarthria: Compensatory and Rehabilitative Approaches, in Motor Speech Disorders, Weismer, (Ed.) San Diego, CA: Plural Publishing, 261-303.
- [Background] Shriberg LD, Aram DM, Kwiatkowski J. Developmental apraxia of speech: III. A subtype marked by inappropriate stress. J Speech Lang Hear Res. 1997 Apr;40(2):313-37. doi: 10.1044/jslhr.4002.313. PMID 9130201
- [Background] Shriberg LD, Lohmeier HL, Strand EA, Jakielski KJ. Encoding, memory, and transcoding deficits in Childhood Apraxia of Speech. Clin Linguist Phon. 2012 May;26(5):445-82. doi: 10.3109/02699206.2012.655841. PMID 22489736
- [Background] Smith A, Goffman L, Zelaznik HN, Ying G, McGillem C. Spatiotemporal stability and patterning of speech movement sequences. Exp Brain Res. 1995;104(3):493-501. doi: 10.1007/BF00231983. PMID 7589300
- [Background] Strand EA. Dynamic Temporal and Tactile Cueing: A Treatment Strategy for Childhood Apraxia of Speech. Am J Speech Lang Pathol. 2020 Feb 7;29(1):30-48. doi: 10.1044/2019_AJSLP-19-0005. Epub 2019 Dec 17. PMID 31846588
- [Background] Strand EA, McCauley RJ, Weigand SD, Stoeckel RE, Baas BS. A motor speech assessment for children with severe speech disorders: reliability and validity evidence. J Speech Lang Hear Res. 2013 Apr;56(2):505-20. doi: 10.1044/1092-4388(2012/12-0094). Epub 2012 Dec 28. PMID 23275421

DOCUMENTS (1):
  • Informed Consent Form (2021-12-01): https://cdn.clinicaltrials.gov/large-docs/53/NCT04642053/ICF_000.pdf